CLINICAL TRIAL: NCT05629650
Title: Effects of 12-week Tai Chi Program on Physical Function, Depression, and Quality of Life Among Cognitively Impaired Older Adults: A Feasibility Study
Brief Title: Feasibility Study of Tai Chi for Cognitively Impaired Older Adults
Acronym: TCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chungnam National University (Other)
Collaborators: National Research Foundation, Singapore (Other Government)
Responsible Party: Principal Investigator, Rhayun Song, Professor, Chungnam National University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ChungnamNU3
Record Dates: First submitted 2022-11-12; First posted 2022-11-29 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Cognitive Impairment
Keywords: Tai Chi; cognitive impairment; dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: two intervention groups (1) those with MCI (2) those with dementia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tai Chi for memory (Experimental): TCM is a standardized type of Tai Chi for health developed by Dr. Lam specifically for those who experience or want to prevent cognitive problems. TCM, consisting of 12 Sun-style and Yang-style Tai Chi movements, can be provided while sitting and while standing with five blocked movement sets so that cognitively impaired individuals (MCI vs. dementia) are able to follow them.
  Interventions: Behavioral: Tai Chi for memory

INTERVENTIONS:
Behavioral: Tai Chi for memory — The adapted form of TCM will be provided at 60 minutes per session, twice a week for 12 weeks by a certified Tai Chi instructor who had experience in teaching older adults with cognitive impairments.

SUMMARY:
The goal of this clinical trial is to determine the feasibility of a 12-week program of Tai Chi for memory (TCM) among older adults with mild cognitive impairment (MCI) or dementia and to determine the effects of TCM on physical functioning, depression, and health-related QoL. Two experimental groups will be recruited for inclusion criteria of community-residing older adults with a diagnosis of either MCI or Dementia.

DETAILED DESCRIPTION:
The purpose of the study are to determine the acceptability of a 12-week program of Tai Chi for memory (TCM) among older adults with mild cognitive impairment (MCI) or dementia; and to determine the effects of TCM on physical functioning, depression, and health-related QoL.

A quasi-experimental design was used with two groups classified according to the level of their cognitive impairment (MCI vs. Dementia).

Depression, health-related QoL, and physical functioning including grip strength, balance, flexibility, and mobility were measured before and after the 12-week TCM program.

Depression was measured using the Korean version of the Geriatric Depression Scale.

Health-related QoL was measured using the 12-item Short Form survey (SF-12). Grip strength was assessed using a digital hand dynamometer. Flexibility was assessed using the standard sit-and-reach test. Balance was measured using the one-leg-standing balance test. Mobility was assessed using the timed up and go test. Paired and independent t-tests will be used to compare the effects of TCM within and between groups.

ELIGIBILITY:
Inclusion Criteria:

* community-residing older adults aged 75 years or older,
* registered at the public dementia prevention centers for dementia screening by health professionals with the diagnosis of either MCI or dementia,
* Korean version of the Montreal Cognitive Assessment (MoCA-K) score of 22 or lower,
* agreed to participate in the Tai Chi program twice a week for 12 weeks.

Exclusion Criteria:

* participated in any formal regular exercise program during the previous 6 months, and

Ages: 75 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
physical function-grip strength | changes from pretest to 12 week posttest scores
  grip strength by assessed in both hands using a digital hand dynamometer (0-90 kg; Labisen KS-301)
physical function - flexibility | changes from pretest to 12 week posttest scores
  by the standard sit-and-reach test (SSRT)
physical function - balance | changes from pretest to 12 week posttest scores
  assessed using a one-leg-standing balance test (OLST)
physical function - mobility | changes from pretest to 12 week posttest scores
  assessed by the Timed Up and Go test (TUG)

SECONDARY OUTCOMES:
emotional functioning - depression | changes from pretest to 12 week posttest scores
  assessed by the short form of the Korean version of the Geriatric Depression Scale (SGDS-K) with 16 items (yes/no). higher scores indicate more depressive symptoms
Short Form Health Survey 12 (SF12) | changes from pretest to 12 week posttest scores
  Short Form Health Survey 12, which consists of eight dimensions: general health, physical functioning, role physical, body pain, vitality, social functioning, role emotional, and mental health. two summary scores for the physical and mental components of health-related QoL are calculated by using the weighted means for the eight domains.

CONTACTS AND LOCATIONS:
Overall Officials: Rhayun Song, PhD, Principal Investigator — Chungnam National University
Locations (1):
- Tai Chi for health institute, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: Yes
upon request, study protocol and the data without individual IDs can be shared with other researchers.
Supporting Information: Study Protocol, CSR
Time Frame: January-December, 2024
Access Criteria: researchers or reviewers who requested for clinical study or meta-analysis

REFERENCES:
- [Derived] Oh H, Song R, Kim SJ. Effects of 12-week Tai Chi program on physical function, depression, and quality of life among cognitively impaired older adults: a feasibility study. BMC Geriatr. 2023 Mar 3;23(1):118. doi: 10.1186/s12877-023-03840-2. PMID 36869290